CLINICAL TRIAL: NCT04882332
Title: Metformin Usage Index and Vitamin B12 Status in Egyptian Type 2 Diabetic Patients : A Case Control Study .
Brief Title: Metformin Usage Index and Vitamin B12 Status in Egyptian Type 2 Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Youssry Helmy, Lecturer of internal medicine, Cairo University
Other Study IDs: N-25-2021
Record Dates: First submitted 2021-04-28; First posted 2021-05-11 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus
Keywords: metformin usage index; vitamin b 12 status; diabetes control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- metformin usage index and vitamin B12 level: Samples for correlation between metformin usage index and vitamin B1 level will be withdrawn from 108 type 2 diabetes patients
  Interventions: Other: sampling for diabetes control parameters; Other: Sampling for vitamin B12 level

INTERVENTIONS:
Other: sampling for diabetes control parameters — Intravenous blood withdrawal for a sample of fasting blood glucose (FBG), 2 hr postprandial blood glucose (2 hr -PPG), fasting lipids {total cholesterol (TC), triglycerides (TAG), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C)}, glycosylated hemoglobin (Hb A1c) ,fasting insulin level and Vitamin B 12 levels
Other: Sampling for vitamin B12 level — Intravenous blood sampling for a sample of vitamin B12 level

SUMMARY:
Current data estimated that 451 million people, (age 18-99 years) suffered from diabetes world wide in 2017, and are expected to rise to 693 million by 2045. Among them, type 2 diabetes mellitus (T2DM) accounts for around 90% of all cases with diabetes.

T2DM is associated with several deterimental microvascular and macrovascular complications (Annani-Akollor ME et al ., 2019) . As such, effective management of the disease is crucial.

The American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD) recommend metformin as the first therapeutic choice for T2DM management with concurrent lifestyle modifications. Reports indicated that metformin improves peripheral insulin sensitivity and reduces the risk of cardiovascular mortality in T2DM in addition to its beneficial effects on weight loss and vascular protection.

Nonetheless, as with most medications, metformin has some side effects. Though most of these side effects are mild, reports indicated that metformin use is associated with diminution of vitamin B12 level . Also, advanced age of patients with T2DM, nutritional deficiency, and malabsorption are other contributing factors for its deficiency .

The proposed mechanisms for deficiency include, impairment of calcium dependent absorption from the gut, alteration in small bowel motility resulting in bacterial overgrowth, and a reduction in intrinsic factor levels .

Metformin-induced vitamin B12 deficiency has also been associated with neuropathy. The neuropathy associated with vitamin B12 deficiency ranges from paresthesia and attenuated peripheral sensation in response to changes in mental status and proprioception which overlap with diabetic neuropathy.

The progression of vitamin B12 deficiency-induced neurologic damage can, however, be abated through early detection and vitamin B12 therapy. Nonetheless, if peripheral neuropathy due to deficiency of vitamin B12 is misconstrued as diabetic peripheral neuropathy , permanent neurological damage may occur.

Several studies have investigated the individual effects of the dose and duration of metformin therapy on vitamin B12 levels .The reported results are inconsistent, with some studies reporting an association with the dose but not the duration and other studies reporting an association only for the duration. however, A few studies did not find an association with either the dose or the duration..

This could be attributed to the fact that, in any given patient with T2DM, vitamin B12 levels could be influenced predominantly by either the dose or the duration of metformin therapy. Hence, it is important to involve both the dose and duration of metformin therapy into the assessment of vitamin B12 deficiency.

Micronutrient deficiencies constitute a global health issue, particularly among countries in the Middle East .The World Health Organization (WHO) has divided this region into overlapping country clusters with regard to nutrition stages and dominant nutrition problems, including major risk factors and underlying causes, program interventions, and gaps in response to these problems.

Countries in early nutrition transition (e.g., Egypt, Jordan, Lebanon, Morocco, and Palestine) are typically characterized by a moderate prevalence of overweight and obesity, moderate levels of undernutrition in specific population groups, and widespread micronutrient deficiencies/inadequacies.

Metformin Usage Index is the product of the dose of metformin (mg) used and its duration divided by 1000. An index which incorporates both of these factors would not only be useful to understand the cumulative impact on vitamin B12 levels but also provide an objective threshold for initiating vitamin B12 supplementation .

So , the aim of this study is to assess the relationship between the dose and duration of metformin therapy with vitamin B12 levels using the "Metformin Usage Index" (MUI) in Egyptian type 2 diabetic patients where the incidence of nutritional deficiencies are not uncommom in order to formulate their appropriate management strategies .

The aim of our study is to evaluate the combined effect of both dose and duration of metformin therapy on vitamin B12 levels in Egyptian patients with type 2 diabetes mellitus (T2D).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 to 65 years old with controlled and uncontrolled type 2 DM

Exclusion Criteria:

* T2DM patients who are pregnant/lactating women,
* newly diagnosed with T2DM (< 3 months),
* who receive vitamin B12 supplementation or proton-pump inhibitors over the last 6 months,
* alcoholics ,
* known cases of malabsorption (gastrointestinal surgery, inflammatory bowel diseases and gluten allergy),
* chronic kidney disease,
* pernicious anemia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 108 patients aged 20 to 65 years old with controlled and uncontrolled type 2 DM
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between Metformin Usage Index and Vitamin B12 status among Egyptian patients with type 2 diabetes | 6 months
  The relationship between MUI and vitamin B12 levels will be assessed among the studied groups

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
not to share

REFERENCES:
- [Background] Ahmed MA, Muntingh G, Rheeder P (2016) Vitamin B12 deficiency in metformin-treated type-2 diabetes patients, prevalence and association with peripheral neuropathy. BMC Pharmacol Toxicol 17(1):44. https ://doi.org/10.1186/s4036 0-016-0088-3. Alvarez M, Sierra OR, Saavedra G, Moreno S (2019) Vitamin B12 deficiency and diabetic neuropathy in patients taking metformin: a cross-sectional study. Endocr Connect 8(10):1324- 1329. https ://doi.org/10.1530/EC-19-0382. Annani-Akollor ME, Addai-Mensah O, Fondjo LA, et al.(2019) Predominant complications of type 2 diabetes in kumasi: a 4-year retrospective cross-sectional study at a teaching hospital in Ghana. Medicina (B Aires). 2019;55(5): 125.